CLINICAL TRIAL: NCT01789138
Title: Randomized Controlled Trial of Situated Optimal Adherence Intervention Estonia (sOAI Estonia) Among Persons Living With HIV/AIDS (PLWHA) on Antiretroviral Therapy (ART) in Estonia
Brief Title: Adherence Support Intervention for Persons Living With HIV/AIDS (PLWHA) on Antiretroviral Therapy (ART) in Estonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Collaborators: National Institute for Health Development, Estonia (Other Government)
Responsible Party: Principal Investigator, Anneli Uusküla, Professor of Epidemiology, Department of Public Health, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SARTH12115T; 3.2.1001.11-0020 (Other Grant/Funding Number: ERDF, Estonian Healthcare Programme, self-funding)
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: HIV; AIDS; Medication Adherence
Keywords: Antiretroviral Therapy; Adherence; Intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Situated Optimal Adherence Intervention (Experimental): Situated Optimal Adherence Intervention: see 'Interventions' for more details.
  Interventions: Behavioral: Situated Optimal Adherence Intervention
- Adherence counseling, standard of care (No Intervention): Standard of care: Antiretroviral therapy adherence is discussed with patient (study participant) according to usual practice in the medical institution no special protocol followed.

INTERVENTIONS:
Behavioral: Situated Optimal Adherence Intervention — Situated Optimal Adherence Intervention consists of 3 individual sessions (during consecutive medication pick-up visits to the clinic) -- patient-centered, non-judgmental, Motivational Interviewing- and theory-based, semi-structured, brief, candid conversations with a trained clinical care nurse using the Next Step Counseling approach. The intervention targets: accurate information about ART (mechanisms of HIV and antiretrovirals) and the development of mental imagery around it; promotion of perceived sense of ease and efficacy in working the ART regimen into the context of one's daily life and circumstances that may challenge drug use persistence; identification and refinement of skills that promote ease of adhering to one's ART regimen across the diverse and challenging contexts.
  Arms: Situated Optimal Adherence Intervention

SUMMARY:
The specific aim of the study is to assess antiretroviral therapy adherence and evaluate the impact of a situated treatment adherence intervention program among persons living with HIV/AIDS on antiretroviral therapy in Estonia.

DETAILED DESCRIPTION:
Specific antiretroviral therapy (ART) can suppress HIV replication and consequently preserve the functioning of immune system. ART is a lifelong treatment with several different concomitantly administered oral medications. According to studies, low adherence to treatment is directly related to knowledge and beliefs about ART.

Studies have shown the success of different interventions increasing adherence to ART, but additional studies need to be carried out in order to determine the most effective components of the interventions and the methods most suitable considering the local context, that could be easily incorporated into the working routine of an medical institution (clinic) with limited extra resources.

Primary locations to implement activities directed at improving treatment adherence are medical institutions, i.e. the departments of infectious diseases where persons living with HIV/AIDS receive their ART.

The aim of the study is to conduct a small-scale intervention (randomised controlled) study implementing a brief adherence counseling targeting persons receiving ART.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* aware of the HIV-positive status for at least 3 months
* ≥ 18 years of age
* speak and read either Estonian or Russian
* receive or start (on recruitment date) antiretroviral therapy

Exclusion Criteria:

* pregnant
* under the influence of alcohol or (illicit)drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Uusküla, MD, MSc, PhD, Principal Investigator — University of Tartu
Locations (2):
- Estonia (2):
  - West-Tallinn Central Hospital, Tallinn, Harju
  - East-Viru Central Hospital, Kohtla-Järve, Ida-Virumaa

IPD SHARING:
Plan to Share IPD: Undecided
Currently considering.

REFERENCES:
- [Background] Chesney MA, Ickovics JR, Chambers DB, Gifford AL, Neidig J, Zwickl B, Wu AW. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committee of the Adult AIDS Clinical Trials Group (AACTG). AIDS Care. 2000 Jun;12(3):255-66. doi: 10.1080/09540120050042891. PMID 10928201
- [Background] R Amico K, McMahan V, Goicochea P, Vargas L, Marcus JL, Grant RM, Liu A. Supporting study product use and accuracy in self-report in the iPrEx study: next step counseling and neutral assessment. AIDS Behav. 2012 Jul;16(5):1243-59. doi: 10.1007/s10461-012-0182-5. PMID 22460228
- [Background] Fisher JD, Amico KR, Fisher WA, Harman JJ. The information-motivation-behavioral skills model of antiretroviral adherence and its applications. Curr HIV/AIDS Rep. 2008 Nov;5(4):193-203. doi: 10.1007/s11904-008-0028-y. PMID 18838059
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Uuskula A, Laisaar KT, Raag M, Smidt J, Semjonova S, Kogan J, Amico KR, Sharma A, Dehovitz J. Antiretroviral therapy (ART) adherence and correlates to nonadherence among people on ART in Estonia. AIDS Care. 2012;24(12):1470-9. doi: 10.1080/09540121.2012.672724. Epub 2012 Apr 25. PMID 22533736
- [Background] Laisaar KT, Avi R, DeHovitz J, Uuskula A. Estonia at the threshold of the fourth decade of the AIDS era in Europe. AIDS Res Hum Retroviruses. 2011 Aug;27(8):841-51. doi: 10.1089/aid.2010.0223. Epub 2011 Jan 11. PMID 21142588

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 519 participants (259 intervention + 260 control arm) randomized. Written informed consent forms of 2 not available (filed). Post-randomization study site control revealed 5 participants not having met the inclusion criterion 'receive or start (on recruitment date) ART'. Data of 512 participants (254 intervention + 258 control arm) analysed.
Period: Overall Study
Arm/Group | Situated Optimal Adherence Intervention | Adherence Counseling, Standard of Care
Started | 254 | 258
Completed | 213 | 206
Not Completed | 41 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Situated Optimal Adherence Intervention | Adherence Counseling, Standard of Care | Total
Number analyzed (Participants) | 254 | 258 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.08 (8.02) | 33.92 (7.65) | 34.00 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 94 | 207
  Male | 141 | 164 | 305
Region of Enrollment [Number; unit: participants]
  Estonia | 254 | 258 | 512
Viral load [Number; unit: participants] — HIV-1 RNA (viral load) with sensitivity of 40 copies/mL.
  participants
    undetectable viral load | 109 | 87 | 196
    detectable viral load | 81 | 91 | 172
    data not available | 64 | 80 | 144
Treatment adherence [Number; unit: participants] — Patient self-reported 3-day recall measure: Counting pills prescribed and taken in past 3 days. Adherent when >=95% of pills taken as prescribed.
  participants
    adherent | 190 | 189 | 379
    non-adherent | 22 | 25 | 47
    data not available | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Antiretroviral Therapy (ART) Adherence (Self-reported 3-day Recall Measure)
Time Frame: 12 months
Population: Number of participants who completed the study
Measure: Number; unit: participants
Arm/Group | Situated Optimal Adherence Intervention | Adherence Counseling, Standard of Care
Number analyzed (Participants) | 213 | 206
participants
  >=95% adherent at baseline and 12 mo | 142 | 139
  >=95% adherent at baseline, but <95% at 12 mo | 6 | 12
  <95% adherent at baseline and 12 mo | 0 | 8
  <95% adherent at baseline, but >=95% at 12 mo | 17 | 8
  data not available (at month 12) | 48 | 39

2. Secondary Outcome: HIV-1 RNA Count / Viral Load (VL)
Description: Undetectable viral load: HIV-1 RNA <40 copies/mL
Time Frame: 12 months
Population: Number of participants who completed the 12-month study
Measure: Number; unit: participants
Arm/Group | Situated Optimal Adherence Intervention | Adherence Counseling, Standard of Care
Number analyzed (Participants) | 213 | 206
participants
  undetectable VL at baseline and 12 mo | 62 | 53
  undetectable VL at baseline, detectable at 12 mo | 7 | 6
  detectable VL at baseline and 12 months | 30 | 37
  detectable VL at baseline, undetectable at 12 mo | 18 | 19
  data not available (at month 12) | 96 | 91

ADVERSE EVENTS:
Arm/Group | Situated Optimal Adherence Intervention | Adherence Counseling, Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/258
Other Adverse Events (participants affected / at risk) | 0/254 | 0/258

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No